CLINICAL TRIAL: NCT07280546
Title: Analysis of Breath Sounds During Surgery
Acronym: BREATHSOUND
Status: Recruiting | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-09-002AC
Record Dates: First submitted 2025-09-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: General Anesthesia; Intraoperative Monitoring; Respiratory Sounds
Keywords: Breath sounds; Perioperative care; Airway monitoring; Respiratory complications; Double-lumen endotracheal tube (DLT)
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation Group: Patients undergoing elective surgery under general anesthesia with endotracheal intubation. Electronic stethoscope patches will be placed to record and analyze intraoperative breath sounds. Target enrollment: 30 participants.
  Interventions: Other: Electronic stethoscope monitoring

INTERVENTIONS:
Other: Electronic stethoscope monitoring — Application of electronic stethoscope patches on the patient's chest during surgery to record breath sounds for subsequent analysis. No therapeutic intervention is given; this is a monitoring/observational tool.

SUMMARY:
This study aims to analyze breath sounds during surgery by using electronic stethoscope sensors attached to patients under general anesthesia. The study will evaluate whether breath sound monitoring can provide useful information for respiratory management, assist anesthesiologists in early detection of abnormal breathing events, and support safer perioperative care. A total of 30 adult patients undergoing elective surgery under general anesthesia will be enrolled.

DETAILED DESCRIPTION:
Continuous breath sound monitoring has the potential to provide anesthesiologists with real-time physiological information that is not captured by standard perioperative monitors. During general anesthesia, subtle changes in airflow or airway patency may precede clinically apparent respiratory compromise. Traditional auscultation is intermittent, subjective, and dependent on the operator's experience. Recent advances in electronic stethoscope technology enable continuous, high-fidelity acquisition of breath sound signals, allowing quantitative analysis and automated detection of abnormal respiratory patterns.

In this prospective observational study, adult patients undergoing elective surgery under general anesthesia will have electronic stethoscope sensors placed on the anterior chest wall prior to induction. Breath sound signals will be continuously recorded throughout anesthesia and surgery. Signal acquisition parameters (sampling rate, filtering, and sensor placement) will be standardized across participants. All breath sound recordings will be synchronized with standard intraoperative monitoring data, including respiratory rate, tidal volume, capnography, pulse oximetry, and hemodynamic parameters. The synchronized dataset will allow temporal correlation between acoustic features and clinically documented respiratory events.

Collected signals will undergo post-processing to extract quantitative acoustic features such as amplitude, frequency distribution, airflow-related patterns, and event-associated spectral changes. Episodes suggestive of abnormal respiration-such as diminished breath sounds, irregular airflow patterns, obstruction-like signatures, or apnea-like silent periods-will be identified and compared with clinical observations recorded by anesthesia providers. The study will also evaluate the feasibility of integrating continuous breath sound information into perioperative workflows, including the practicality of sensor placement, stability of recordings during surgical manipulation, and compatibility with existing monitoring systems.

The overall goal of the study is to generate foundational evidence on the technical feasibility and clinical relevance of continuous breath sound monitoring under general anesthesia. Findings from this study may support future development of automated respiratory event detection tools and may contribute to safer perioperative respiratory management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for elective surgery under general anesthesia
* Provided written informed consent

Exclusion Criteria:

* History of respiratory disease (e.g., COPD, severe asthma)
* Previous airway surgery or anatomical abnormalities that interfere with breath sound assessment
* Refusal to participate or inability to comply with study procedures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult surgical patients (aged 20 years or older) scheduled for elective surgery under general anesthesia at Taipei Veterans General Hospital, Taiwan. Eligible patients are ASA I-III and willing to provide informed consent. Patients with significant respiratory disease or airway abnormalities will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of electronic breath sound monitoring during surgery | During surgery (from induction of anesthesia until emergence)
  Assessment will be based on the proportion of intraoperative respiratory events correctly identified by the electronic breath sound monitoring system compared with standard clinical assessment.

SECONDARY OUTCOMES:
Incidence of respiratory events detected by the device | Intraoperative period.
  Number of intraoperative respiratory events (e.g., hypoventilation, airway obstruction, disconnection) identified by the monitoring system.
Correlation between electronic breath sound monitoring and clinical observation | Intraoperative period.
  Correlation (r-value) between device output and anesthesiologist-documented respiratory findings.
User feasibility and device performance | Immediately after surgery (postoperative evaluation).
  Feasibility will be assessed by reporting the proportion of cases in which continuous breath sound monitoring was successfully completed without interruption, including documentation of signal quality issues and workflow interference if present. (No rating scale will be used.)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsuan Ke, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified breath sound recordings and corresponding clinical parameters (e.g., age, ASA physical status, type of anesthesia) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available starting 6 months after study completion and for up to 5 years.
Access Criteria: Qualified researchers who provide a methodologically sound research proposal and obtain approval from an independent ethics committee/IRB may request access to de-identified individual participant data (IPD). Requests should be directed to the Institutional Review Board (IRB) of Taipei Veterans General Hospital, Taiwan. Data will be shared through secure platforms to ensure confidentiality and compliance with ethical regulations.
URL: https://clinicaltrials.gov

REFERENCES:
- [Background] Manecke GR Jr, Dilger JP, Kutner LJ, Poppers PJ. Auscultation revisited: the waveform and spectral characteristics of breath sounds during general anesthesia. Int J Clin Monit Comput. 1997 Nov;14(4):231-40. doi: 10.1007/BF03356568. PMID 9451573
- [Background] Mansy HA, O'Connor CJ, Balk RA, Sandler RH. Breath sound changes associated with malpositioned endotracheal tubes. Med Biol Eng Comput. 2005 Mar;43(2):206-11. doi: 10.1007/BF02345956. PMID 15865129
- [Background] Wei TJ, Hsiung PY, Liu JH, Lin TC, Kuo FT, Wu CY. Use of Electronic Auscultation in Full Personal Protective Equipment to Detect Ventilation Status in Selective Lung Ventilation: A Randomized Controlled Trial. Front Med (Lausanne). 2022 Feb 21;9:851395. doi: 10.3389/fmed.2022.851395. eCollection 2022. PMID 35265648
- See also: Institutional Review Board of Taipei Veterans General Hospital — https://wd.vghtpe.gov.tw/irb/Index.action
- See also: Frontiers in Medicine - Electronic Auscultation Trial — https://doi.org/10.3389/fmed.2022.851395
- Available data/document: Study Protocol — https://www.vghtpe.gov.tw/Index.action — The study protocol describing the methodology of electronic auscultation of breath sounds during anesthesia will be available. De-identified respiratory sound data and related analysis scripts may be shared upon reasonable request to the principal investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Full Protocol and SAP (Version 1.0)_1206 (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT07280546/Prot_SAP_000.pdf